CLINICAL TRIAL: NCT05845957
Title: The Efficiency of Education Given to Students With Digital Storytelling in Safe Pediatric Intravenous Drug Administration
Brief Title: Digital Storytelling in Pediatric Safe Drug
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Şeyda BİNAY YAZ, Assistant professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bakircay
Record Dates: First submitted 2023-04-17; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Education; Nursing; Innovativeness
Keywords: Nursing students; Education; Digital stroytelling; pediatrics; safe drug application

STUDY DESIGN:
Intervention Model Description: The research was a randomized controlled, experimental study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Education Group (Experimental): All participants in this group were given the "Safe pediatric intravenous drug administration knowledge test" prepared by the researchers as a pre-test.
  The participants of this group, who were determined by randomization, were given training prepared using the digital storytelling method. The training took 25 minutes.
  After the training, the "Safe intravenous drug administration knowledge test" was applied as a post-test.
  Interventions: Other: Digital Education Group
- Control Group (No Intervention): No intervention was made. All participants in this group were given the "Safe pediatric intravenous drug administration knowledge test" prepared by the researchers as a pre-test.
  Afterward, theoretical information on the subject was given. After theoretical information, the "Safe intravenous drug administration knowledge test" was applied as a post-test.

INTERVENTIONS:
Other: Digital Education Group — Providing training on safe pediatric intravenous drug administration with digital storytelling method
  Arms: Digital Education Group

SUMMARY:
Summary Aim: This research was conducted to determine the effectiveness of education given to students using digital storytelling in safe pediatric intravenous drug administration.

Method: It is a randomized controlled experimental study. The sample of the study consisted of 84 nursing students. The students included in the study were divided into two equal groups: the experimental and control groups. Digital education material of the experimental group and theoretical education was applied to the control group. Before and after the training, a post-knowledge test was made and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of the Department of Nursing
* Taking the child health and diseases nursing course and being successful
* Volunteering to participate in the research

Exclusion Criteria:

* Participate and quit the study
* Being a 1st and 2nd year nursing student
* Failure of the child health and diseases nursing course

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Statistical difference between groups about knowledge test scores | During the education, approximately 25 minutes
  Safe pediatric drug practices knowledge test is applied twice as pre-test and post-test in experimental and control groups.
  Safe pediatric drug practices knowledge test: It is a 17-question form prepared by researchers. Content validity has been made for the form. Each correct answer is calculated as 1 point and each wrong answer is calculated as 0 points. The higher the score obtained from the questionnaire, the higher the level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Akkoyun, Principal Investigator — Izmir Bakircay University
Locations (1):
- Semih, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be prepared for publication